CLINICAL TRIAL: NCT05759299
Title: International obServational sTudy on AiRway manaGement in operAting Room and Non-operaTing Room anaEsthesia
Acronym: STARGATE
Status: Recruiting | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: STARGATE
Record Dates: First submitted 2023-02-24; First posted 2023-03-08 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Airway Complication of Anesthesia
Keywords: airway management; anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing anesthesia in operating room and outside operating room: Patients undergoing elective or emergency advanced airway management to receive general anesthesia for surgery in operating room or outside operating room (e.g. endoscopy and radiology unit, cardiology lab cath)
  Interventions: Procedure: Advanced airway management

INTERVENTIONS:
Procedure: Advanced airway management — Advanced airway management with either tracheal intubation or supraglottic airways performed after induction with hypnotic and/or opioid drugs

SUMMARY:
According to WHO, more than 230 million major surgical procedures are carried out under general anaesthesia each year worldwide. Despite important technological advances, airway management remains a major challenge in anaesthesiology. Data from large perspective studies on current incidence of major peri-intubation adverse events are lacking in the anaesthesia setting, especially on outcomes such as peri-intubation cardiovascular collapse, severe hypoxemia, and cardiac arrest. These events are more common in case of difficulties with airway management so that first pass intubation failure significantly increase the risks. Moreover, it has been documented that even transient hypotension during general anaesthesia, may have long-term consequences and may be associated with a worse outcome in patients undergoing non-cardiac surgery. The primary aim of the study is to assess the current incidence of major adverse events during advanced airway management for anaesthesia in patients undergoing elective or emergency surgery and in the setting of nonoperating room anesthesia. The secondary aim is to assess the current practice of airway management during anesthesia worldwide.

STARGATE Study will be a large international observational study recruiting all consecutive adult (≥ 18 years old) patients undergoing general anesthesia in operating room and outside operating room. Primary outcome will be a composite of cardiovascular collapse, cardiac arrest and severe hypoxemia.

DETAILED DESCRIPTION:
According to WHO, more than 230 million major surgical procedures are carried out under general anaesthesia each year worldwide. Despite important technological advances, airway management remains a major challenge in anesthesiology. Data from large perspective studies on current incidence of major peri-intubation adverse events are lacking in the anesthesia setting, especially on outcomes such as peri-intubation cardiovascular collapse, severe hypoxemia, and cardiac arrest. These events are more common in case of difficulties with airway management so that first pass intubation failure significantly increase the risks. Moreover, it has been documented that even transient hypotension during general anesthesia, may have long-term consequences and may be associated with a worse outcome in patients undergoing non-cardiac surgery. The primary aim of the study is to assess the current incidence of major adverse events during advanced airway management for anesthesia in patients undergoing elective or emergency surgery and in the setting of non-operating room anesthesia. The secondary aim is to assess the current practice of airway management during anesthesia worldwide.

Study design: International, multicenter, prospective cohort study

Inclusion criteria: We will include all adult (≥ 18 years old) patients undergoing advanced airway management for general anaesthesia in operating room (OR) or non-operating room anaesthesia (NORA).

Exclusion criteria: Airway management during cardiopulmonary resuscitation; critically ill patients undergoing intubation due to their underlying clinical condition.

Primary outcome: At least one of the following major peri-intubation adverse events occurring within 30 minutes from induction or up to surgical incision: severe hypoxia, cardiovascular collapse, cardiac arrest.

Study duration: All centers will enroll all consecutive patients meeting study criteria up to 50 maximum patients for each center.

Collected data: We will collect the following information:

* Informed consent and admission data
* Demographic and clinical characteristics
* Type of procedure (time, setting, type of surgery, elective or emergency
* Airway evaluation (anticipated difficult airway management)
* Monitoring applied during the procedure
* Patient's parameters
* Preoxygenation method and use of apnoeic oxygenation (position during preoxygenation, rapid sequence induction applied)
* Drugs used for induction (molecules and doses)
* Elective method for laryngoscopy
* Operator's characteristics
* Method used for the second (and following) attempt
* Method used for adequate tube placement confirmation
* Duration of laryngoscopy
* Outcome of endotracheal intubation (total number of attempts, laryngoscopy view, minimum SpO2 during laryngoscopy, need for LMA)
* Intubation-related complications (severe cardiovascular collapse, severe and mild hypoxemia, cardiac arrest, airway injury or any bleeding, aspiration of gastric contents, dental injury, emergency front of neck airway (FONA), cannot intubate cannot oxygenate scenario (CICO), unplanned need for ICU secondary to airway management complications)
* Extubation procedure.

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥ 18 years old) patients undergoing advanced airway management for general anaesthesia in operating room (OR) or non-operating room anaesthesia (NORA).

Exclusion Criteria:

* Airway management during cardiopulmonary resuscitation.
* Critically ill patients undergoing intubation due to their underlying clinical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, not critically ill patients, undergoing advanced airway management (i.e. tracheal intubation or supraglottic airways) to receive surgery or any kind of diagnostic or therapeutic procedure under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 10500 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Major peri-intubation adverse event | 30 minutes from induction
  Defined as at least one of the following events:
  * Cardiovascular collapse (at least one of the following):
    1. Systolic arterial pressure < 65 mmHg
    2. Systolic arterial pressure < 90 mmHg for > 15 minutes
    3. New need of vasopressors and/or fluid load > 15 ml/kg to maintain the target blood pressure
  * Cardiac arrest
  * Severe hypoxemia (SpO2 < 80%)

SECONDARY OUTCOMES:
Minor peri-intubation adverse events | 30 minutes from induction
  At least one of the following:
  * Moderate hypoxia (SpO2 < 93%)
  * Airway injury
  * Clinically relevant bleeding
  * Oral aspiration of gastric contents
  * Dental injury
Difficult facemask ventilation | 30 minutes from induction
  Impossibility to provide adequate ventilation because of one or more of the following problems: inadequate mask seal, excessive gas leak, or excessive resistance to the ingress or egress of gas
First pass success rate | 30 minutes from induction
  Incidence of successful intubation after a single attempt of laryngoscopy

OTHER OUTCOMES:
Emergency front of neck access (eFONA) | 30 minutes from induction
  Emergency need for invasive access to the patient's neck to provide adequate oxygenation (e.g. cricothyroidotomy, percutaneous tracheostomy, surgical tracheostomy).
Cannot intubate cannot oxygenate (CICO) | 30 minutes from induction
  Impossibility to achieve a successful tracheal intubation and adequate patient's oxygenation
Unplanned need for ICU secondary to airway management complications | 24 hours from induction
  Unplanned admission to ICU after an airway-related complication or prolonged/difficult instrumentation
In-hospital mortality | 28 days from induction
  Death during the same hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Russotto, MD, Principal Investigator — University of Turin, Italy; Francesca Collino, MD, Principal Investigator — University of Turin, Italy
Locations (10):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Cochin University Hospital, Assistance Publique - Hôpitaux de Paris, Paris, France
- Tata Memorial Hospital, Mumbai, India
- University Hospital of Galway, Galway, Ireland
- Italy (5):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza E Brianza
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano, TO
  - A.O.U. Città della Salute e della Scienza, Torino, TO
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale Santa Chiara, APSS Trento, Trento

REFERENCES:
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Background] Cook TM. Strategies for the prevention of airway complications - a narrative review. Anaesthesia. 2018 Jan;73(1):93-111. doi: 10.1111/anae.14123. PMID 29210033
- [Background] Russotto V, Myatra SN, Laffey JG, Tassistro E, Antolini L, Bauer P, Lascarrou JB, Szuldrzynski K, Camporota L, Pelosi P, Sorbello M, Higgs A, Greif R, Putensen C, Agvald-Ohman C, Chalkias A, Bokums K, Brewster D, Rossi E, Fumagalli R, Pesenti A, Foti G, Bellani G; INTUBE Study Investigators. Intubation Practices and Adverse Peri-intubation Events in Critically Ill Patients From 29 Countries. JAMA. 2021 Mar 23;325(12):1164-1172. doi: 10.1001/jama.2021.1727. PMID 33755076
- [Background] Russotto V, Tassistro E, Myatra SN, Parotto M, Antolini L, Bauer P, Lascarrou JB, Szuldrzynski K, Camporota L, Putensen C, Pelosi P, Sorbello M, Higgs A, Greif R, Pesenti A, Valsecchi MG, Fumagalli R, Foti G, Bellani G, Laffey JG. Peri-intubation Cardiovascular Collapse in Patients Who Are Critically Ill: Insights from the INTUBE Study. Am J Respir Crit Care Med. 2022 Aug 15;206(4):449-458. doi: 10.1164/rccm.202111-2575OC. PMID 35536310
- [Background] Green RS, Erdogan M. Are outcomes worse in patients who develop post-intubation hypotension? CJEM. 2022 Aug;24(5):465-466. doi: 10.1007/s43678-022-00340-x. Epub 2022 Aug 2. No abstract available. PMID 35917027
- [Background] Green RS, Butler MB. Postintubation Hypotension in General Anesthesia: A Retrospective Analysis. J Intensive Care Med. 2016 Dec;31(10):667-675. doi: 10.1177/0885066615597198. Epub 2016 Jul 7. PMID 26721639
- [Background] Apfelbaum JL, Hagberg CA, Connis RT, Abdelmalak BB, Agarkar M, Dutton RP, Fiadjoe JE, Greif R, Klock PA, Mercier D, Myatra SN, O'Sullivan EP, Rosenblatt WH, Sorbello M, Tung A. 2022 American Society of Anesthesiologists Practice Guidelines for Management of the Difficult Airway. Anesthesiology. 2022 Jan 1;136(1):31-81. doi: 10.1097/ALN.0000000000004002. PMID 34762729
- [Background] Cook TM, MacDougall-Davis SR. Complications and failure of airway management. Br J Anaesth. 2012 Dec;109 Suppl 1:i68-i85. doi: 10.1093/bja/aes393. PMID 23242753
- [Background] Rose DK, Cohen MM. The incidence of airway problems depends on the definition used. Can J Anaesth. 1996 Jan;43(1):30-4. doi: 10.1007/BF03015954. PMID 8665631
- [Background] Sudfeld S, Brechnitz S, Wagner JY, Reese PC, Pinnschmidt HO, Reuter DA, Saugel B. Post-induction hypotension and early intraoperative hypotension associated with general anaesthesia. Br J Anaesth. 2017 Jul 1;119(1):57-64. doi: 10.1093/bja/aex127. PMID 28974066
- [Derived] Russotto V, Sansovini C, Muraccini M, Collino F, Myatra SN, Higgs A, Brewster D, Curic Radivojevic R, Parotto M, Karamchandani K, Landoni G, Sorbello M, Monfroglio M, Rovescala G, Martinelli P, Tinelli O, Meessen J, Bellani G, Laffey JG, Langeron O, Caironi P. Multicentre international observational study on airway management for anaesthesia: the STARGATE study protocol. BMJ Open. 2026 Feb 6;16(2):e109038. doi: 10.1136/bmjopen-2025-109038. PMID 41651535